CLINICAL TRIAL: NCT02334683
Title: Comparison of Electrophysiologic And Ultrasound Guidance For Onabotulinum Toxin A Injections in Focal Upper Extremity Dystonia And Spasticity
Brief Title: Compare Two Guidance Techniques for Botulinum Toxin Injections for the Treatment of Limb Spasticity and Focal Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, David M. Simpson, Professor of Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: GCO 14-1113; #86127 (Other: Allergan Pharmaceuticals Funding Agency); NCT02326818 (obsolete NCT alias)
Record Dates: First submitted 2014-12-24; First posted 2015-01-08 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Spasticity; Focal Dystonia; Tremor, Limb
Keywords: Comparison; Botulinum toxin treatments; Ultrasound; Electrophysiologic; Spasticity; Focal dystonia
MeSH Terms: conditions — Muscle Spasticity; Dystonic Disorders; Tremor | interventions — Electric Stimulation; Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrophysiologic guidance (Experimental): Electrophysiologic guidance, using electrical stimulation
  Interventions: Device: Electrical stimulation
- Ultrasound guidance (Active Comparator): Ultrasound guidance,using sound waves through a wand directed towards the targeted muscles.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Electrical stimulation — The purpose of this study is to investigate the use of two ways of locating the muscle for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity located by either electrical stimulation using a needle or ultrasound using sound waves.
  Other Names: E-stim
  Arms: Electrophysiologic guidance
Device: Ultrasound — The purpose of this study is to compare how the muscle is located by either electrical stimulation using a needle or ultrasound using sound waves.
  Other Names: Sonography
  Arms: Ultrasound guidance

SUMMARY:
This study seeks to compare the use of ultrasound and electrophysiologic techniques to target muscles for the treatment of spasticity and focal dystonia of the limbs. The purpose of this study is to investigate the use of two ways of locating the muscle for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity. Electrophysiologic guidance, using electrical stimulation, and ultrasound are the standard ways of locating muscles during a treatment of BoNT injection.

DETAILED DESCRIPTION:
This is a study to investigate the use of two targeting techniques for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity: Electrophysiologic guidance, using electrical stimulation, and ultrasound. Subjects will be selected from the clinical programs of both Icahn School of Medicine at Mount Sinai and the National Institutes of Health who are already receiving onabotulinum toxin A injections clinically. The study will consist of four visits. Visit one consists of screening subjects who will then be consented and randomized to one of the two treatment techniques for their ona-BoNT injection: 1) Electrophysiologic guidance using electrical stimulation or 2) ultrasound. Visit 2 will occur at week 4 where the subjects will return for a follow up visit to have blinded evaluator measurements of efficacy and strength and capture safety data. Visit 3 will be at week 12 when subjects will cross over and have the alternate treatment technique during their ona-BoNT injection. Visit 4 will occur at week 16 as the final assessment where subjects will have measurements of efficacy and strength and capture safety data by the blinded evaluator.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Confirmed diagnosis of focal upper extremity dystonia (FHD) or upper limb spasticity
* Stable onabotulinumtoxinA dose regimen with a stable response as judged by the physician and patient for at least 2 treatment sessions.

Exclusion Criteria:

* Contraindications to botulinum toxin
* Pregnancy or nursing
* Cognitive impairment that prevents reliable outcome measures of self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simpson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Ninds, Nih, Bethesda, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrophysiologic Guidance Then Ultrasound Guidance: Electrophysiologic guidance, using electrical stimulation to locate the muscle for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity located by either electrical stimulation using a needle.
  Ultrasound guidance, using sound waves through a wand directed towards the targeted muscles.
- Ultrasound Guidance Then Electrophysiologic Guidance: Ultrasound guidance, using sound waves through a wand directed towards the targeted muscles.
  Electrophysiologic guidance, using electrical stimulation to locate the muscle for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity located by either electrical stimulation using a needle.
Period: First 12 Week Period
Arm/Group | Electrophysiologic Guidance Then Ultrasound Guidance | Ultrasound Guidance Then Electrophysiologic Guidance
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second 12 Week Period
Arm/Group | Electrophysiologic Guidance Then Ultrasound Guidance | Ultrasound Guidance Then Electrophysiologic Guidance
Started | 9 | 10
Completed | 9 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was done only on the participants who completed at least one cycle - 1 subject from MSSM was lost to follow and is not included
Groups:
- Electrophysiologic Guidance Then Ultrasound Guidance: Electrophysiologic guidance, using electrical stimulation
  Electrical stimulation: The purpose of this study is to investigate the use of two ways of locating the muscle for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity located by either electrical stimulation using a needle or ultrasound using sound waves.
  Ultrasound guidance,using sound waves through a wand directed towards the targeted muscles.
  Ultrasound: The purpose of this study is to compare how the muscle is located by either electrical stimulation using a needle or ultrasound using sound waves.
- Ultrasound Guidance Then Electrophysiologic Guidance: Ultrasound guidance,using sound waves through a wand directed towards the targeted muscles.
  Ultrasound: The purpose of this study is to compare how the muscle is located by either electrical stimulation using a needle or ultrasound using sound waves.
  Electrophysiologic guidance, using electrical stimulation
  Electrical stimulation: The purpose of this study is to investigate the use of two ways of locating the muscle for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity located by either electrical stimulation using a needle or ultrasound using sound waves.
- Total: Total of all reporting groups
Arm/Group | Electrophysiologic Guidance Then Ultrasound Guidance | Ultrasound Guidance Then Electrophysiologic Guidance | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (15.4) | 59.7 (10.8) | 57.53 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 5 | 8 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 10 | 19
  Not Hispanic or Latino | 9 | 10 | 19
Diagnosis [Count of Participants; unit: Participants]
  Spasticity | 5 | 6 | 11
  Dystonia | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Global Impression of Change
Description: clinical or patient self-rating form for grading evaluation of the treatment at 16 weeks as compared to at 4 weeks.
  Full scale from 0 = no improvement and 100 normal use. Higher score indicates better health outcome.
Time Frame: 4 weeks and 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Electrophysiologic Guidance: Electrical stimulation: the use of two ways of locating the muscle for botulinum toxin (BoNT) injection for the treatment of focal hand dystonia and upper limb spasticity located by electrical stimulation using a needle .
- Ultrasound Guidance: Ultrasound guidance, using sound waves through a wand directed towards the targeted muscles.
Arm/Group | Electrophysiologic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 18 | 19
score on a scale | 53.1 [40.2 to 66.0] | 51.5 [38.9 to 64.0]

2. Secondary Outcome: Change in Visual Analog Scale
Description: patient perception of satisfaction and comfort at 16 weeks as compared to at 4 weeks.
  Full scale from 0 = no improvement to 100 = normal. Higher score indicates more improvement.
Time Frame: 4 weeks and 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrophysiologic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 18 | 19
score on a scale | 54.72 (32.21) | 52.37 (31.36)

3. Secondary Outcome: Change in Muscle Strength
Description: Muscle strength measured by dynamometry at 16 weeks as compared to at 4 weeks.
  Full scale 0 = no weakness and 100 is unable to move. Higher score indicates poorer health outcome.
Time Frame: 4 weeks and 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrophysiologic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 18 | 19
score on a scale | 29.89 (27.78) | 20.63 (28.27)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Analysis was done only on the participants who completed at least one cycle - 1 subject from MSSM was lost to follow and is not included
Arm/Group | Electrophysiologic Guidance | Ultrasound Guidance
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electrophysiologic Guidance (N=19) | Ultrasound Guidance (N=19)
Severe Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT02334683/Prot_SAP_000.pdf